CLINICAL TRIAL: NCT03545906
Title: Telemedicine Enhanced Asthma Management - Uniting Providers
Acronym: TEAM-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: University of Arkansas (Other); University at Buffalo (Other)
Responsible Party: Principal Investigator, Jill Halterman, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 72009
Record Dates: First submitted 2018-05-17; First posted 2018-06-04 (Actual); Results first posted 2025-09-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Asthma in Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAM-UP Intervention Group (Experimental)
  Interventions: Other: TEAM-UP Intervention Group
- Enhanced Care Comparison Group (Active Comparator)
  Interventions: Other: Enhanced Care Comparison

INTERVENTIONS:
Other: TEAM-UP Intervention Group — Children randomly assigned to TEAM-UP will have a telemedicine assisted specialist visit scheduled after 4 weeks of initiating DOT at school, as well as 2 subsequent follow-up visits. The visits will be performed by a specialist in pediatric asthma, to implement guideline-based care. Prescriptions for asthma medications will be prescribed to be delivered as directly observed therapy in school.
  Arms: TEAM-UP Intervention Group
Other: Enhanced Care Comparison — Similar to the TEAM-UP group, children in the Enhanced Care group will receive a symptom assessment and asthma education materials at baseline, and we will contact the PCP by facsimile or email and will recommend DOT of preventive asthma medication through school as well as a referral to specialist. However specialist visits will not be facilitated via telemedicine.
  Arms: Enhanced Care Comparison Group

SUMMARY:
This research study is an innovative school-based program for urban children with moderate to severe persistent or difficult-to-control asthma. The Telemedicine Enhanced Asthma Management-Uniting Providers (TEAM-UP) program enhances a school-based, primary care directed asthma program with specialist-supported care to ensure optimal guideline based treatment. This study is a full-scale randomized trial of TEAM-UP versus an enhanced care comparison group. Primary care physicians (PCP) of all enrolled children (n=360, 4-12 yrs.) will be prompted to initiate directly observed therapy (DOT) of preventive asthma medication through school and to make a specialist referral. For children in the TEAM-UP group, the specialist visits will be facilitated via telemedicine at school. The telemedicine specialist visit will be scheduled after approximately 4 weeks of initiating DOT, in order to allow for accurate guideline-based assessments of medication and care needs once adherence with a daily controller medication is established. There will also be up to 2 telemedicine follow-up specialist visits to assess the child's response to treatment and make needed adjustments. The study will use the existing community infrastructure by implementing both telemedicine and DOT in school, and maintaining collaboration with PCPs. Blinded follow-ups will occur at 3-, 5-, 7- and 12-months after baseline, and the primary outcome is the comparison of symptom-free days (SFD) at each follow-up time point.

ELIGIBILITY:
Inclusion Criteria:

1. Physician-diagnosed asthma (based on parent report with validation from the child's physician).
2. Age >=4 and =<12 years.
3. Residence in the City of Rochester and surrounding suburbs, with a. primary residence within the following zip codes: 14445, 14604, 14605, 14606, 14607, 14608, 14609, 14610, 14611, 14612, 14613, 14614, 14615, 14616, 14617, 14618, 14619, 14620, 14621, 14622, 14623, 14624, 14625, 14626.
4. Moderate-severe persistent severity (requiring Step 3 or higher care) or difficult to control asthma despite therapy (based on age-specific NHLBI guidelines).

Exclusion Criteria:

1. Inability to speak and understand English or Spanish. (*Parents unable to read will be eligible, and all instruments will be given verbally.)
2. Current participation in an asthma study.
3. Planning to leave the Rochester city school district area in fewer than 6 months.
4. Having received asthma specialist care in the prior 3 months.
5. Having other significant medical conditions, including congenital heart disease, cystic fibrosis, or other chronic lung disease, that could interfere with the assessment of asthma-related measures.
6. In foster care or other situations in which consent cannot be obtained from a guardian.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 326 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2025-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Halterman JS, Fagnano M, Tremblay PJ, Perry TT, Wang H, Mustafa SS, Ramsey A, Stern J. Effect of the Telemedicine Enhanced Asthma Management-Uniting Providers (TEAM-UP) Program on Asthma Outcomes: A Randomized Clinical Trial. J Pediatr. 2025 Oct 23;289:114872. doi: 10.1016/j.jpeds.2025.114872. Online ahead of print. PMID 41139012

RESULTS

PARTICIPANT FLOW:
Groups:
- TEAM-UP Intervention Group: TEAM-UP Intervention Group: Children randomly assigned to TEAM-UP will have a telemedicine assisted specialist visit scheduled after approximately 4 weeks of initiating DOT at school, as well as up to 2 subsequent follow-up visits. The visits will be performed by a specialist in pediatric asthma, to implement guideline-based care. Prescriptions for asthma medications will be prescribed to be delivered as directly observed therapy in school.
Period: Overall Study
Arm/Group | TEAM-UP Intervention Group | Enhanced Care Comparison Group
Started | 163 | 163
Completed | 139 | 137
Not Completed | 24 | 26

BASELINE CHARACTERISTICS:
Population: There was one participant randomized to the TEAM-UP intervention. Shortly after the baseline assessment, it was discovered that the participant did not meet enrollment criteria and was withdrawn from the study. This participant's data is not included in the outcomes.
Groups:
- Total: Total of all reporting groups
Arm/Group | TEAM-UP Intervention Group | Enhanced Care Comparison Group | Total
Number analyzed (Participants) | 162 | 163 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (2.3) | 8.5 (2.5) | 8.35 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 68 | 130
  Male | 100 | 95 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 59 | 113
  Not Hispanic or Latino | 108 | 104 | 212
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 96 | 91 | 187
  White | 8 | 9 | 17
  More than one race | 22 | 28 | 50
  Unknown or Not Reported | 36 | 34 | 70
Region of Enrollment [Number; unit: participants]
  United States | 162 | 163 | 325
Public Insurance [Count of Participants; unit: Participants] | 128 | 132 | 260
Symptom-free days over 2 weeks [Mean (Standard Deviation); unit: days] | 6.36 (5.1) | 6.84 (5.3) | 6.6 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Mean Symptom-Free Days in Prior 14 Days
Description: Mean number of symptom-free days in the prior 14 days (range 0-14)
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TEAM-UP Intervention Group | Enhanced Care Comparison Group
Number analyzed (Participants) | 154 | 149
days | 9.21 (4.8) | 8.21 (5.0)
Statistical Analysis 1: Comparison: TEAM-UP Intervention Group vs Enhanced Care Comparison Group; Test type: Superiority; p = .075, t-test, 2 sided; Mean Difference (Net) = 1

2. Primary Outcome: Mean Symptom-Free Days in Prior 14 Days
Description: Mean number of symptom-free days in the prior 14 days (range 0-14)
Time Frame: 5 months after baseline
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TEAM-UP Intervention Group | Enhanced Care Comparison Group
Number analyzed (Participants) | 147 | 150
days | 10.4 (4.5) | 9.1 (4.8)
Statistical Analysis 1: Comparison: TEAM-UP Intervention Group vs Enhanced Care Comparison Group; Test type: Superiority; p = .018, t-test, 2 sided; Mean Difference (Net) = 1.3

3. Primary Outcome: Mean Symptom-Free Days in Prior 14 Days
Description: Mean number of symptom-free days in the prior 14 days (range 0-14)
Time Frame: 7 months after baseline
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TEAM-UP Intervention Group | Enhanced Care Comparison Group
Number analyzed (Participants) | 143 | 142
days | 10.1 (4.9) | 8.9 (5.0)
Statistical Analysis 1: Comparison: TEAM-UP Intervention Group vs Enhanced Care Comparison Group; Test type: Superiority; p = .039, t-test, 2 sided; Mean Difference (Net) = 1.2

4. Primary Outcome: Mean Symptom-Free Days in Prior 14 Days
Description: Mean number of symptom-free days in the prior 14 days (range 0-14)
Time Frame: 12 months after baseline
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TEAM-UP Intervention Group | Enhanced Care Comparison Group
Number analyzed (Participants) | 139 | 137
days | 9.6 (5.1) | 8.9 (5.4)
Statistical Analysis 1: Comparison: TEAM-UP Intervention Group vs Enhanced Care Comparison Group; Test type: Superiority; p = .265, t-test, 2 sided; Mean Difference (Net) = .7

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | TEAM-UP Intervention Group | Enhanced Care Comparison Group
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/163
Serious Adverse Events (participants affected / at risk) | 12/163 | 10/163
Other Adverse Events (participants affected / at risk) | 0/163 | 0/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEAM-UP Intervention Group (N=163) | Enhanced Care Comparison Group (N=163)
Hospitalizations due to asthma (Respiratory, thoracic and mediastinal disorders) | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT03545906/Prot_SAP_000.pdf